CLINICAL TRIAL: NCT05300347
Title: Prospective Observational Study Evaluating the Prevalence of Adenosine Deaminase (ADA) Enzyme Deficiency Disease in Adult Patients With Bronchiectasis, Lymphopenia and/or Immunoglobulin E Elevation in Pulmonology Clinics
Brief Title: Observational Study Evaluating the Prevalence of Enzyme Deficiency in Pulmonology Clinics (ADA)
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: TRPHARM (Industry)
Responsible Party: Sponsor
Other Study IDs: TR-ADA-005
Record Dates: First submitted 2022-03-18; First posted 2022-03-29 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Bronchiectasis; Adenosine Deaminase Deficiency; Pulmonary Disease
Keywords: lymphopenic, Immunoglobulin E, bronchiectasis
MeSH Terms: conditions — Bronchiectasis; Severe combined immunodeficiency due to adenosine deaminase deficiency; Lung Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: adenosine deaminase enzyme deficiency test — adenosine deaminase enzyme deficiency

SUMMARY:
This observational study was designed as a prospective epidemiological screening study. Patients who applied to the centers participating in the study, bronchiectasis was detected on at least one computed tomography of the lungs; Immunoglobulin E height and/or were found to be lymphopenic on at least one examination will be included in the study. Up-to-date data will be collected from patients who have agreed to participate in the study, and a blood sample with DBS will be taken from patients. The blood taken will be subjected to analysis for ADA metabolites. For patients with a high metabolic test, the responsible researcher will advise on clarifying the diagnosis with a genetic test other than the study. In case of formation of new information for each patient, consultation will be provided by the responsible researcher. Thus, the prevalence of ADA enzyme deficiency disease in patients with bronchiectasis, Immunoglobulin E elevation and/or lymphopenia will be evaluated. In addition, with this study, it will be scientifically demonstrated whether lymphopenia and/or Immunoglobulin E height is a parameter that facilitates the early diagnosis of patients with late-onset ADA enzyme deficiency.

DETAILED DESCRIPTION:
Bronchiectasis is a chronic disease characterized by abnormal and persistent expansion of the bronchi. Although its frequency is not clearly known in our country, it is considered to be 53-566/100,000 in the Guidelines of the European Society of Respiratory Diseases. Of genetic origin (cystic fibrosis, Primary ciliary dyskinesia, etc.), as well as recurrent lung infections (pneumonia,viral infections, etc.) it can also develop depending on. Bronchiectasis due to recurrent lung infections may occur in patients with primary immunodeficiency. Primary immunodeficiency diseases are a group of diseases that are accompanied by chronic and/or recurrent bacterial, fungal, protozoal and viral infections that develop as a result of primary or congenital immunodeficiency. The incidence dec in society varies from 1/10,000 to 1/100,000. Combined immunodeficiencies account for 15-29% of primary immunodeficiencies. Severe Combined Immuno Deficiencies (SCID) are a heterogeneous group of diseases caused by hereditary errors in genes involved in the development and/or function of T, B, and sometimes NK cells, which cause serious dysfunction of the immune system. The incidence is estimated at 1/100,000 live births in the United States. Although the exact incidence of inbreeding is not known in our country, where inbreeding is common, it is expected that those who show autosomal recessive transition will be more common, especially. The recognition of these disorders by clinicians is important for reducing long-term complications due to recurrent infections and preventing mortality with appropriate treatment. The frequency of SCID in our country is unknown. Unlike in Europe and America, SCID types, which are autosomal recessive in our country, are considered to be the most common form due to high rates of inbreeding. The number obtained by comparing the number of live babies born in a year in Konya with the number of AKIY cases diagnosed in the Pediatric Immunology clinic of the Meram Faculty of Medicine of Selcuk University, the only primary immunodeficiency diagnostic center in the region, in the same year, is 1/10,000. This preliminary study shows that in our country this disease is much more common than in Europe and America. To date, more than 20 genetic defects that cause SCID have been identified. All known genetic defects disrupt the development of cells of the immune system, causing combined immunodeficiency. One of them, the ADA defect, is also a metabolic disease, due to which there is a lack of enzymes. ADA catalyzes the deamination of purine nucleosides adenosine (Ado) and 2'-deoxyadenosine (dAdo), which are produced during the degradation and transformation of RNA and DNA. ADA is a cleansing enzyme; it detoxifies purines. In ADA deficiency, 2'-deoxyadenosine (dAdo) is phosphorylated and converted into deoxyadenosine triphosphate (dATP). Accumulation of DATP disrupts DNA repair and replication. A high percentage of dATP accumulates in ADA deficiency, especially in erythrocytes and lymphocytes. Increased levels of adenosine break down the wall of the lymphocyte. It inhibits the development of lymphocytes in the thymus. A kind of lymphocyte intoxication occurs. It leads to a severe form of lymphopenia. Approximately 10-20% of AKIS are diagnosed as ADA enzyme deficiency. It shows an autosomal recessive transition. Your gene is 20. it is localized on the long arm of the chromosome. Clinically, there are early and late onset types.

Classic-early onset ADA deficiency: Although normal at birth, patients present with infections seen from the first months of life, resulting in death if left untreated. In addition to the AKI table, neuro-developmental disorders, sensorineural hearing loss and/or skeletal abnormalities have also been reported in these patients. Although hematopoietic stem cell transplantation, enzyme replacement therapy and gene therapy are treatment approaches that provide cure, early diagnosis determines the prognosis.

Late onset ADA deficiency: Patients may present with recurrent infections, bronchiectasis, autoimmunity, human papilloma virus (HPV) infections at an older age, even in adulthood. Lymphopenia is an invariable finding. High IgE and eosinophilia may be observed. In these cases, residual enzyme activity due to the type of mutation causes a late onset. This phenotype accounts for 10-15% of all cases of ADA deficiency. Patients with late-onset ADA enzyme deficiency appear in the form of case reports. in a study conducted in Zurich in 1997, where the data of two patients were shared, it was observed that one patient had a history of recurrent otitis and pulmonary infection, bronchiectasis, lymphopenia, and immunoglobulin E elevation. The other patient, his cousin ADA, was diagnosed by chance while undergoing a bone marrow scan due to enzyme deficiency. There is a history of recurrent tonsillitis. in a study conducted by Hacettepe University published in 2018, the data of 13 patients with ADA enzyme deficiency were evaluated, and 3 patients with late/delayed diagnosis were found to have ADA enzyme deficiency. A patient with a late diagnosis of ADA enzyme deficiency was found to have recurrent pneumonia, bronchiectasis, and Immunoglobulin E elevation. In the study in which the data of a patient with a late onset ADA enzyme deficiency published in Konya from our country in 2010 were shared, it was observed that the patient had a history of resection of the lower left lobe due to bronchiectasis, lymphopenia and immunoglobulin E elevation.

Diagnosis: ADA enzyme deficiency is included in severe combined immunodeficiencies and is observed with lymphopenia and infections. The diagnosis is made by measuring the activity of the enzyme ADA in erythrocytes or lymphocytes in patients with suspected clinical and laboratory features (such as lymphopenia, bronchiectasis). By mutation analysis, a gene defect is shown. However, T-cell receptor excision circles (TREC) test is used for early diagnosis. However, since the TREC test is found to be normal at birth in late-onset patients, screening that leads patients to an early diagnosis can only be achieved by measuring ADA metabolites. In late-onset ADA deficiency, it is difficult to diagnose. Low awareness of the disease and its symptoms usually results in these cases not being diagnosed, not being able to reach effective treatment, permanent organ damage and patient loss. For this reason, diagnosis of patients is very important in terms of quality of life, as well as vital importance. Reasons: ADA enzyme deficiencies account for approximately 15% of severe combined immunodeficiencies. 15-20% of patients with ADA enzyme deficiency have a late diagnosis of ADA enzyme deficiency. Because of the inability of these patients to get a diagnosis, their treatment is also inadequate. This is the first time in our country.

the aim of the study is to investigate the ADA metabolites in the target group of adult patients with bronchiectasis, lymphopenia and/or Immunoglobulin E elevation by looking at the diagnosis and to obtain preliminary data on the prevalence of ADA disease.

ELIGIBILITY:
Inclusion Criteria:

Signing of the written informed consent form by the patient and/or his legal representative,

* Detection of bronchiectasis (cystic fibrosis, non-primary ciliary dyskinesia) on at least one computed tomography of the patient's lungs,
* The patient is between dec8 and 40 years of age.
* Patients with at least one major and one minor criteria from the following criteria will be included in the study:

Major Criteria:

1. Lymphopenia: lymphopenia as a result of at least one hemogram of the patient exist,

   -The number of lymphocytes is below 1500/mm3
2. Immunoglobulin E height: 120 kU/L of immunoglobulin E level having it on

Minor Criteria:

1. Two or more new ear infections within a year
2. Two or more new sinus infections within a year when there is no allergy
3. One pneumonia per year for more than a year
4. Chronic diarrhea with weight loss
5. Recurrent viral infections (Colds, herpes, warts, condyloma)
6. The need for repeated intravenous antibiotics to clear infections
7. Recurrent deep skin or internal organ abscesses
8. Persistent thrush or fungal infection of the skin or other place
9. Infection caused by tuberculosis-like bacteria that is normally harmless
10. Primary immunodeficiency in the family

Exclusion Criteria:

1. The patient was diagnosed with ADA enzyme deficiency before being included in the study,
2. Congenital bronchiectasis before inclusion in the study (cystic fibrosis, primary ciliary dyskinesia,alpha-1 anti trypsin deficiency, etc. diagnosed,
3. Having used drugs that may cause lymphopenia before being included in the study (chemotherapy, cytotoxic drug use, etc.),
4. The Ministry of Health COVID-19 diagnosis guide (nazofaringeal, nasal orofaringiyal or SARS-CoV-2 RNA PCR test and/or tomographic) as COVID-19, diagnosed and/or persons who had contact with patients diagnosed in this manner, even karsilasal patient recruitment criteria, these patients will be taken after PCR tests were negative in the study.
5. Before being included in the study, it should be noted that other diseases that can cause lymphopenia (hematological diseases, oncological diseases, etc.) have been diagnosed with,
6. The patient has participated in an interventional clinical trial within the last 30 days,
7. Conclusion-In the opinion of the researcher, the patient will not be able to properly fulfill the study requirements,
8. Pregnancy-the period of pregnancy and/or lactation,
9. The fact that the volunteer participating in the study received an erythrocyte suspension or a complete blood transfusion within the last 3 months.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: male and female patients between the ages of 18 and 40
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2021-06-17 (Actual); Primary Completion 2021-09-23 (Actual); Study Completion 2023-06-17 (Estimated)

PRIMARY OUTCOMES:
It is the determination of the prevalence of ADA enzyme deficiency | 2 years
  Bronchiectasis is the determination of the prevalence of ADA enzyme deficiency disease in adult patients with Immunoglobulin E elevation and/or lymphopenia.

SECONDARY OUTCOMES:
Determination of late-onset ADA enzyme deficiency | 2 years
  Determination of clinical and laboratory characteristics of late-onset ADA enzyme deficiencies

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara University Medical Faculty, Ankara, Mamak, Turkey (Türkiye)